CLINICAL TRIAL: NCT06465589
Title: PRIVATE - Preference Research: Investigating Variations of Anonymity, Transparency, and Efficacy in Digital Health Applications
Brief Title: Variations of Anonymity, Transparency, and Efficacy in Digital Health Applications
Acronym: PRIVATE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-00842; 10002000 (Other: University of Bern, Department of Clinical Psychology and Psychotherapy, internal ID); SNCTP000005924 (Registry Identifier: Swiss National Clinical Trials Portal (SNCTP))
Record Dates: First submitted 2024-06-13; First posted 2024-06-20 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Social Anxiety
Keywords: Social Anxiety; Mental Disorders; Internet Intervention; Self Help; Preference
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: The study is a single-center partially randomized patient preference trial with four conditions (program version: standard vs. anonymous and allocation: randomized vs. preferred)
Who Masked: Investigator
Masking Description: The investigators will not know which specific condition the participants were in for the initial analysis. The blind will be broken for the investigators after first interpretation of the results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Randomized Anonymous (Experimental): After participants are randomized to the randomization arm, they will once again be randomized to the program versions. Participants in this arm will use the anonymous program.
  Interventions: Other: JOURNeY anonymous
- Randomized Standard (Active Comparator): After participants are randomized to the randomization arm, they will once again be randomized to the program versions. Participants in this arm will use the standard program.
  Interventions: Other: JOURNeY standard
- Preferred Anonymous (Other): After participants are randomized to the preference arm, they will be given access to the program version they indicate a preference for after having read two descriptive texts about both versions. Participants in this arm will use the anonymous program.
  Interventions: Other: JOURNeY anonymous
- Preferred Standard (Other): After participants are randomized to the preference arm, they will be given access to the program version they indicate a preference for after having read two descriptive texts about both versions. Participants in this arm will use the standard program.
  Interventions: Other: JOURNeY standard

INTERVENTIONS:
Other: JOURNeY anonymous — The anonymously usable version of the self-help program JOURNeY which does not require a login and does not collect personal data.
  Includes 4 main components:
  1. psychoeducation where participants learn about SAD and the treatment,
  2. cognitive restructuring where participants challenge dysfunctional social cognitions,
  3. attention training where participants learn to decrease self-focused attention, and
  4. exposure where participants seek out and endure fear-inducing situations.
  Additionally, there is a first module which discusses motivation and a conclusion module which encourages participants to keep practicing and using techniques they learned in the program in their daily life.
  Arms: Preferred Anonymous; Randomized Anonymous
Other: JOURNeY standard — The standard version of the self-help program JOURNeY which requires a login and collects personal data.
  Includes 4 main components:
  1. psychoeducation where participants learn about SAD and the treatment,
  2. cognitive restructuring where participants challenge dysfunctional social cognitions,
  3. attention training where participants learn to decrease self-focused attention, and
  4. exposure where participants seek out and endure fear-inducing situations.
  Additionally, there is a first module which discusses motivation and a conclusion module which encourages participants to keep practicing and using techniques they learned in the program in their daily life.
  Arms: Preferred Standard; Randomized Standard

SUMMARY:
Social Anxiety Disorder (SAD) is one of the most widespread mental illnesses and it has previously been shown that online therapy and online self-help tools such as the one investigated in this study can be successful in reducing not only symptoms of SAD but also symptoms of depression and increase the quality of life of participants. A substantial concern with digital health intervention tools is data security and privacy as many such tools have been found to be unsafe and easy targets for hacker attacks, potentially endangering personal (health) data of the users.

For this research project, an internet-based program targeting social anxiety has been developed that can be used completely anonymously (i.e., without collecting an email address or other information that can or could potentially identify users). This new anonymized version will be compared in a partially randomized patient preference trial with an already well-evaluated version in which, as is common in other digital health applications, personal data such as the email address or other information from the users is used, for example, for login.

Study objectives:

1. To investigate the efficacy of a completely anonymous version of the program "JOURNeY" based on cognitive behavioral therapy (CBT) and compare it to an already evidence-based non-anonymous version of the program regarding primary social anxiety symptoms, and secondary outcomes such as depressive symptoms, quality of life, usability, adherence to the program, internalized stigma, attitudes on help-seeking, and personality functioning.
2. To investigate patients' preferences and the influence of patients' preferences on outcome.
3. To explore how patient characteristics are associated with participants' preferences.

DETAILED DESCRIPTION:
Social Anxiety Disorder (SAD) is one of the most widespread mental illnesses and it has previously been shown that online therapy and online self-help tools such as the one investigated in this study can be successful in reducing not only symptoms of SAD but also symptoms of depression and increase the quality of life of participants. A substantial concern with digital health intervention tools is data security and privacy as many such tools have been found to be unsafe and easy targets for hacker attacks, potentially endangering personal (health) data of the users.

For this research project, an internet-based program targeting social anxiety has been developed that can be used completely anonymously (i.e., without collecting an email address or other information that can or could potentially identify users). It is originally based on the well-established cognitive-behavioral treatment of social anxiety by Clark and Wells from 1995. This new anonymized version will be compared in a partially randomized patient preference trial with an already well-evaluated version in which, as is common in other digital health applications, personal data such as the email address or other information from the users is used, for example, for login. The fully anonymized version has some disadvantages regarding usability and possibly also effectiveness, as no usage history can be stored, users cannot pick up where they left off during a new login, and instead of entering texts in diaries, for example, about anxiety-related thoughts within the program, they need to download a PDF, etc. On the other hand, the anonymized version has advantages regarding the low threshold for use and privacy. People who could benefit from such internet-based programs might be more likely to use them, as there are no data protection risks associated with their use, and a fully anonymized version could immediately be used even without entering an email address. Thus, the reach and impact of evidence-based digital tools for mental problems and disorders such as social anxiety (disorder) could be increased with an anonymous version. However, there are no studies on the effectiveness of digital tools which can be used anonymously and there is no knowledge about the preferences of users (e.g., is it important for users to be able to use an anonymous version, or do they prefer the non-anonymized version with a few practical advantages?).

Study objectives:

1. To investigate the efficacy of a completely anonymous version of the CBT-based program "JOURNeY" and compare it to an already evidence-based non-anonymous version of the program regarding primary social anxiety symptoms, and secondary outcomes such as depressive symptoms, quality of life, usability, adherence to the program, internalized stigma, attitudes on help-seeking, and personality functioning.
2. To investigate patients' preferences and the influence of patients' preferences on outcome.
3. To explore how patient characteristics are associated with participants' preferences.

This study is part of a larger trial conducted with two departments at the University of Bern. One part assesses clinical research questions and the other part is concerned with psychology of digitalization which researches user behavior and concerns regarding privacy in digital health applications.

The study is a single-center partially randomized patient preference trial and for the clinical part, there are two experimental factors (program versions, i.e. anonymous and standard) each evaluated at two levels (randomized vs. preferred).

Recruitment: Participants will be recruited using reports in newspapers, through internet forums, social media (e.g., Facebook), and via a website (https://www.online-therapy.ch/) in German-speaking countries.

Sampling: After checking the inclusion criteria, participants will be randomized with equal probability to one of the two conditions; randomization vs. preference. In the second stage, if a participant is randomized to the choice arm, the participant can choose the preferred treatment; if a participant is randomized to the random arm, the participant is randomized to a program version (anonymous vs. standard) arm. This design is used to estimate the treatment, selection, and preference effect. The random allocation will be unknown to the investigators. In order to keep the sample sizes of the 16 conditions similar, the allocation list will be made using randomly permuted blocks.

A total of 452 participants who exceed pre-defined cut-off scores on social anxiety measures will be recruited for this study.

Assessment procedures: The primary outcome measure is change in symptoms of SAD at post-treatment, i.e., after 8 weeks. Secondary outcomes include sustaining change at follow up (6 months after baseline), changes in depressive symptoms, changes in quality of life, changes in internalized stigma and attitudes towards help-seeking, changes in levels of personality functioning, and negative effects. Furthermore, an exploratory preference analysis will be conducted to gain insights into digital health application users' preferences and potential preference effect.

Treatment: The internet-based self-help program ("JOURNeY") is based on the well-established cognitive-behavioral treatment of social anxiety by Clark and Wells from 1995 and has been proven efficacious in previous studies. The standard version of JOURNeY is accessed through a secure website, with each participant having a password-protected account. It consists of the following four treatment components: (1) psychoeducation (knowledge about SAD and its treatment); (2) cognitive restructuring (challenging dysfunctional social cognitions); (3) attention training (decrease of self-focused attention); and (4) exposure (decrease of avoidance of feared situations and safety behaviors). The anonymous version has the same content but does not require an account and does not collect any personal data of participants.

Data analysis: Primary analyses will be conducted on the Intention-To-Treat (ITT) sample (i.e., all assigned participants) using linear mixed models with repeated measures. In addition, a completers analysis will be carried out, also with linear mixed models with repeated measures.

For the preference analysis, a more exploratory approach will be used. For binary outcome data (e.g. program preference), regression analysis will be conducted. For other data, tests such as t-test, chi-squared tests or other appropriate tests will be used.

Reporting will follow CONSORT E-Health standards.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Be 18 years or older,
* Have access to the internet
* Have access to a smartphone, computer or tablet
* Score 22 points or higher on the Social Phobia Scale or 33 points or higher on the Social Interaction Anxiety Scale (SPS & SIAS)

Exclusion Criteria:

* Score 2 points or higher on the suicide item of the PHQ-9
* Have previously been diagnosed with psychotic symptoms or bipolar disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2024-09-03 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Social Anxiety Symptoms | at baseline, 8 Weeks
  Change from baseline in the composite score of two self-report social anxiety questionnaires measuring various symptoms from time pre to time post (Social Phobia Scale & Social Interaction Anxiety Scale; SPS & SIAS). The scales contain a total of 40 items resulting in scores of 0 to 160 with higher scores indicating more severe social anxiety symptoms. The composite score will be the averaged z-score of both questionnaires.

SECONDARY OUTCOMES:
Social Anxiety Symptoms | at baseline, at 8 weeks, at 24 weeks
  Change in the composite score and individual scores of two self-report social anxiety questionnaires measuring various symptoms from time pre to time post and follow-up (Social Phobia Scale & Social Interaction Anxiety Scale; SPS & SIAS). The scales contain a total of 40 items resulting in scores of 0 to 160 with higher scores indicating more severe social anxiety symptoms. The composite score will be the averaged z-score of both questionnaires.
Depressive Symptoms | at baseline, at 8 weeks, at 24 weeks
  Changes in depressive symptoms measured with one self-report questionnaire from time pre to time post and follow-up (Patient Health Questionnaire; PHQ-9). This nine item questionnaire results in scores ranging from 0 to 27 with higher scores indicating more severe depressive symptoms.
Quality of Life QoL | at baseline, at 8 weeks, at 24 weeks
  Changes in quality of Life measured with one self-report questionnaire from time pre to time post and follow-up (Short-Form Health Survey SF-12; SF-12). The twelve items measure quality of life on the two subscales physical and mental aspects. Scores range from 0 to 100 with higher scores indicating higher quality of life.
Internalized Stigma | at baseline, at 8 weeks, at 24 weeks
  Changes in internalized stigma of mental illnesses measured with one self-report questionnaire from time pre to time post and follow-up (Internalized Stigma of Mental Illness Scale; ISMI). It has 29 items and measures stigma on the five subscales alienation, stereotype endorsement, discrimination experience, social withdrawal, and stigma resistance. Overall scores range from 29 to 116 with higher scores indicating higher internalized stigma.
Attitudes Towards Help-Seeking | at baseline, at 8 weeks, at 24 weeks
  Changes of attitudes towards seeking mental health services measured with one self-report questionnaire from time pre to time post and follow-up (Inventory of Attitudes Towards Seeking Mental Health Services; IASMHS). The questionnaire has 24 items with the three subscales psychological openness, help-seeking propensity, and indifference to stigma. Scores range from 0 to 20 for each subscale. For psychological openness and help seeking propensity, higher scores indicate more positive attitudes towards help-seeking. For stigma indifference, higher scores indicate less concern about stigma associated with help-seeking.
Personality Functioning | at baseline, at 8 weeks, at 24 weeks
  Changes in personality functioning measured with one self-report questionnaire from time pre to time post and follow-up (Level of Personality Functioning Scale-Brief Form 2.0; LPFS-BF). This 12-item questionnaire measures personality functioning with the two domains self (subscales: identity and self-direction) and interpersonal (subscales: empathy and intimacy) functioning. Overall scores range from 12 to 48 with higher scores indicating more severe impairment in personality functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Berger, Prof. Dr., Principal Investigator — University Bern, Clinical Psychology and Psychotherapy Department
Locations (1):
- University Bern, Clinical Psychology and Psychotherapy Department, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Clark, D. M., & Wells, A. (1995). A cognitive model of social phobia. In R. G. Heimberg, M. R. Liebowitz, D. Hope, & F. Schneider (Eds.), Social Phobia: Diagnosis, Assessment, and Treatment (pp. 69-93). Guilford Press.
- [Background] Schulz A, Stolz T, Vincent A, Krieger T, Andersson G, Berger T. A sorrow shared is a sorrow halved? A three-arm randomized controlled trial comparing internet-based clinician-guided individual versus group treatment for social anxiety disorder. Behav Res Ther. 2016 Sep;84:14-26. doi: 10.1016/j.brat.2016.07.001. Epub 2016 Jul 7. PMID 27423374
- [Background] Sibitz I, Friedrich ME, Unger A, Bachmann A, Benesch T, Amering M. [Internalized Stigma of Schizophrenia: Validation of the German Version of the Internalized Stigma of Mental Illness-Scale (ISMI)]. Psychiatr Prax. 2013 Mar;40(2):83-91. doi: 10.1055/s-0032-1332878. Epub 2013 Jan 25. German. PMID 23354628
- [Background] Stolz T, Schulz A, Krieger T, Vincent A, Urech A, Moser C, Westermann S, Berger T. A mobile app for social anxiety disorder: A three-arm randomized controlled trial comparing mobile and PC-based guided self-help interventions. J Consult Clin Psychol. 2018 Jun;86(6):493-504. doi: 10.1037/ccp0000301. PMID 29781648
- [Background] Gräfe, K., Zipfel, S., Herzog, W., & Löwe, B. (2004). Screening psychischer Störungen mit dem "Gesundheitsfragebogen für Patienten (PHQ-D)". Diagnostica, 50(4), 171-181. https://doi.org/10.1026/0012-1924.50.4.171
- [Background] Berger T, Caspar F, Richardson R, Kneubuhler B, Sutter D, Andersson G. Internet-based treatment of social phobia: a randomized controlled trial comparing unguided with two types of guided self-help. Behav Res Ther. 2011 Mar;49(3):158-69. doi: 10.1016/j.brat.2010.12.007. Epub 2011 Jan 1. PMID 21255767
- [Background] Kessler EM, Agines S, Bowen CE. Attitudes towards seeking mental health services among older adults: personal and contextual correlates. Aging Ment Health. 2015;19(2):182-91. doi: 10.1080/13607863.2014.920300. Epub 2014 Jun 5. PMID 24898327
- [Background] Wolfangel, E. (2023, May 9). Datenschutz: Wenn Hacker mit Gesundheits-Apps besonders leichtes Spiel haben. ZEIT ONLINE. https://www.zeit.de/digital/datenschutz/2023-05/gesundheitsapp-datenschutz-depression-edupression-sicherheitsluecke/komplettansicht
- [Background] Gandek B, Ware JE, Aaronson NK, Apolone G, Bjorner JB, Brazier JE, Bullinger M, Kaasa S, Leplege A, Prieto L, Sullivan M. Cross-validation of item selection and scoring for the SF-12 Health Survey in nine countries: results from the IQOLA Project. International Quality of Life Assessment. J Clin Epidemiol. 1998 Nov;51(11):1171-8. doi: 10.1016/s0895-4356(98)00109-7. PMID 9817135
- [Background] Batterham P, Gulliver A, Sunderland M, Farrer L, Kay-Lambkin F, Trias A, Calear A. Factors Influencing Community Participation in Internet Interventions Compared With Research Trials: Observational Study in a Nationally Representative Adult Cohort. J Med Internet Res. 2023 Feb 2;25:e41663. doi: 10.2196/41663. PMID 36729613
- [Background] Spitzer C, Muller S, Kerber A, Hutsebaut J, Brahler E, Zimmermann J. [The German Version of the Level of Personality Functioning Scale-Brief Form 2.0 (LPFS-BF): Latent Structure, Convergent Validity and Norm Values in the General Population]. Psychother Psychosom Med Psychol. 2021 Jul;71(7):284-293. doi: 10.1055/a-1343-2396. Epub 2021 Mar 10. German. PMID 33694153
- [Background] Stein DJ, Lim CCW, Roest AM, de Jonge P, Aguilar-Gaxiola S, Al-Hamzawi A, Alonso J, Benjet C, Bromet EJ, Bruffaerts R, de Girolamo G, Florescu S, Gureje O, Haro JM, Harris MG, He Y, Hinkov H, Horiguchi I, Hu C, Karam A, Karam EG, Lee S, Lepine JP, Navarro-Mateu F, Pennell BE, Piazza M, Posada-Villa J, Ten Have M, Torres Y, Viana MC, Wojtyniak B, Xavier M, Kessler RC, Scott KM; WHO World Mental Health Survey Collaborators. The cross-national epidemiology of social anxiety disorder: Data from the World Mental Health Survey Initiative. BMC Med. 2017 Jul 31;15(1):143. doi: 10.1186/s12916-017-0889-2. PMID 28756776
- [Background] Mattick RP, Clarke JC. Development and validation of measures of social phobia scrutiny fear and social interaction anxiety. Behav Res Ther. 1998 Apr;36(4):455-70. doi: 10.1016/s0005-7967(97)10031-6. PMID 9670605
- [Background] Spitzer RL, Kroenke K, Williams JB. Validation and utility of a self-report version of PRIME-MD: the PHQ primary care study. Primary Care Evaluation of Mental Disorders. Patient Health Questionnaire. JAMA. 1999 Nov 10;282(18):1737-44. doi: 10.1001/jama.282.18.1737. PMID 10568646
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Ritsher JB, Otilingam PG, Grajales M. Internalized stigma of mental illness: psychometric properties of a new measure. Psychiatry Res. 2003 Nov 1;121(1):31-49. doi: 10.1016/j.psychres.2003.08.008. PMID 14572622
- [Background] Mackenzie, C. S., Knox, V. J., Gekoski, W. L., & Macaulay, H. L. (2004). An Adaptation and Extension of the Attitudes Toward Seeking Professional Psychological Help Scale1. Journal of Applied Social Psychology, 34(11), 2410-2433. https://doi.org/10.1111/j.1559-1816.2004.tb01984.x
- [Background] Hutsebaut J, Feenstra DJ, Kamphuis JH. Development and Preliminary Psychometric Evaluation of a Brief Self-Report Questionnaire for the Assessment of the DSM-5 level of Personality Functioning Scale: The LPFS Brief Form (LPFS-BF). Personal Disord. 2016 Apr;7(2):192-7. doi: 10.1037/per0000159. Epub 2015 Nov 23. PMID 26595344
- [Background] Weekers LC, Hutsebaut J, Kamphuis JH. The Level of Personality Functioning Scale-Brief Form 2.0: Update of a brief instrument for assessing level of personality functioning. Personal Ment Health. 2019 Feb;13(1):3-14. doi: 10.1002/pmh.1434. Epub 2018 Sep 19. PMID 30230242
- [Derived] Arnold S, Vogt MF, Boettcher J, Fenski F, Sipka D, Elson M, Berger T. A Freely Accessible, Anonymous Online Treatment for Social Anxiety: Protocol for a Partially Randomized Patient Preference Trial. JMIR Res Protoc. 2025 Nov 5;14:e77573. doi: 10.2196/77573. PMID 41192825
- See also: Link to Study Description on Homepage of University of Bern — https://www.dig.psy.unibe.ch/research/current_projects/private_preference_research_investigating_variations_of_anonymity_transparency_and_efficacy/index_eng.html